CLINICAL TRIAL: NCT04331353
Title: Comparative Effectiveness of Multi Versus Single Intervention Allergen Reduction Strategies on Asthma Morbidity
Brief Title: The Allergen Reduction and Child Health Study (ARCHS)
Acronym: ARCHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Felicia Rabito, Associate Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-2199; AD-2018C3-14869 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children
Keywords: asthma; cockroach allergen; indoor allergens; pulmonary function; childhood asthma; environmental intervention
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparator 1 (tailored approach) (Active Comparator): Multi-component intervention tailored to the participant's allergic profile.
  Interventions: Behavioral: Comparator 1 (tailored approach)
- Comparator 2 (insecticidal bait) (Active Comparator): Insecticidal bait for cockroach reduction.
  Interventions: Behavioral: Comparator 2 (insecticidal bait)

INTERVENTIONS:
Behavioral: Comparator 1 (tailored approach) — Tailored to a child's sensitization status. Components include, education, cockroach baiting, mattress and bed covers, high efficiency particulate air (HEPA) vacuum cleaner, air purifier.
  Arms: Comparator 1 (tailored approach)
Behavioral: Comparator 2 (insecticidal bait) — Cockroach bait
  Arms: Comparator 2 (insecticidal bait)

SUMMARY:
The Allergen Reduction and Child Health Study (ARCHS) is a 12-month, two group randomized control trial of children with asthma and who are exposed to cockroaches. Children ages 5 - 17 living in the Greater New Orleans area will be recruited from a variety of clinic and community settings. The overall goal of the study is to improve patient-centered asthma outcomes (asthma symptom days, health care utilization, asthma control and quality of life) by targeting one key allergen - cockroach exposure in the child's home. The investigators propose a simple intervention of insecticidal bait that is low cost, simple to implement, and which is lower toxicity than other forms of pest control. The reduction in the number of cockroaches in the home is an environmental outcome that is patient-centered and is likely to add to its acceptance by families of children with asthma.

DETAILED DESCRIPTION:
Background and Significance: Asthma is a serious, complex, and highly prevalent childhood respiratory disorder leading to inflammation and narrowing of the airways. If uncontrolled it negatively impacts long-term lung function. An estimated 6.2 million, 1 in 12, U.S. children have asthma and asthma outcome disparities are pervasive. An important contributor to asthma disparities is greater exposure to asthma triggering allergens. The proposed study addresses an evidence gap related to the most effective way to reduce exposure to asthma triggers in the home.

Study Aims: There are three specific aims. First to compare the effectiveness of a multicomponent intervention to reduce asthma triggers to a single intervention to reduce cockroach exposure in the home testing the hypothesis that among children with asthma exposed to cockroaches, a single intervention targeting cockroach remediation is as effective one with multiple components that targets multiple allergens. Specific Aim 2 compares the effectiveness of the different interventions on the number of cockroaches in the home testing the hypothesis that insecticidal bait is as effective at reducing cockroaches as a multi-component approach. Specific Aim 3 examines whether the effect of insecticidal control on asthma outcomes differs by the allergen profile of the child. The investigators hypothesize that cockroach eradication results in improved outcomes independent of cockroach sensitization status and the number of other allergens to which a child is sensitized. The long term objective is to provide evidence for the NHLBI Expert Panel currently reviewing the Guidelines for the Diagnosis and Management of Asthma (EPR-3) and specifically the effectiveness of indoor allergen reduction strategies on asthma management.

Study Description: A 12-month, two group randomized clinical trial of 290 children ages 5 -17 with doctor diagnosed asthma recruited from clinics in the Greater New Orleans area. Comparator Group 1 targets dust mites, mold, cockroach, animal dander and smoke exposure. Interventions include asthma education, cleaning techniques, impermeable bed covers, HEPA vacuum cleaners, air purification, and insecticidal baiting. Comparator Group 2 targets cockroaches and the intervention is targeted insecticidal baiting.

Primary outcomes include asthma symptom days, asthma-related health care utilization (emergency room visits, hospitalization, unscheduled clinic visits), quality of life, asthma control, medication use, and cockroach burden. Pulmonary function will be measured as a secondary outcome. Asthma outcome data will be collected monthly. Other data will be collected during home visits at baseline, 3, 6, 9 and 12 months.

Each outcome will be modeled separately. Two sets of analyses will be conducted. First, a generalized linear regression model will be employed to model the change score from baseline to 12-months with Comparator group 2 as the predictor and other potential confounders as covariates. In the second approach, intervention effects will be assessed longitudinally by modelling the outcomes at each assessment time (excluding baseline) using models for repeated outcomes such as linear mixed model or generalized estimating equations depending on the distribution of the outcome. Sensitivity analyses will be performed to verify the stability of multiple imputation assumptions using different multiple imputation procedures and consistency of the final results.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 - 17 years; with uncontrolled persistent asthma defined as the child experiencing at least one of the following: one overnight hospitalization for asthma within the past six months OR two unscheduled clinic or emergency department visits for asthma within the last 12 months; and either on a long term controller medication for asthma, or have asthma symptoms 3 or more days per week over the past 2 weeks or nighttime asthma symptoms at least 3 times in the past month exposure to cockroach - defined as trapping at least one cockroach in a 3 day period OR visual evidence of cockroaches by field staff; and the child must sleep in the target home at least 4 nights per week on average. Caregiver ability to speak English or Spanish.

Exclusion Criteria:

* Other serious medical or chronic illnesses including chronic respiratory infections that require daily medication, cardiovascular disease that requires daily medication, excluding hypertension, taking a beta-blocker, a current active smoker, currently receiving immunotherapy or plans to move within the 12 month follow-up.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum number of symptom days in the previous two weeks | 12 Months
  The number of days with asthma symptoms (chest tightness, cough, wheeze, disrupted sleep, limitations on physical activities) in the previous two weeks.
Number of participants with an asthma related hospitalization, unscheduled clinic or emergency room visit for asthma in the previous month | 12 Months
  Hospitalization or emergency room visit for asthma or unscheduled doctor visit for asthma in the previous month.
Level of Asthma control | 12 Months
  The level of asthma control assessed using the Asthma Control Test. The scores range from 5 to 25 with higher scores reflecting greater asthma control.

SECONDARY OUTCOMES:
Asthma quality of life | 12 Months
  Quality of life measured using the Pediatric Asthma Quality of Life Questionnaire. 7 point Likert scale (Minimum:1 Maximum:7) all items are weighted equally. Higher scores indicate higher quality of life.
Cockroach exposure | Baseline, 3, 6, 9, 12 months
  The number of cockroaches in the home and the level of cockroach antigen in the dust

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Rabito, PhD, Principal Investigator — Tulane University School of Public Health and Tropical Medicine
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No